CLINICAL TRIAL: NCT00866580
Title: Immunogenicity and Safety of GSK Biologicals' (Pre-) Pandemic Influenza Candidate Vaccine GSK 1562902A.
Brief Title: A Study for Evaluation of GSK Biologicals' Pandemic Influenza Vaccine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was cancelled before enrolment for reasons not related to vaccine safety or efficacy.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 112865
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Influenza
Keywords: Pandemic influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: GSK's candidate influenza vaccine 1562902A; Biological: FluarixTM; Biological: Placebo
- Group B (Experimental)
  Interventions: Biological: GSK's candidate influenza vaccine 1562902A; Biological: FluarixTM; Biological: Placebo

INTERVENTIONS:
Biological: GSK's candidate influenza vaccine 1562902A — Intramuscular dose on Day 0 and Day 21
Biological: FluarixTM — Intramuscular dose on Day 42 or on Day -30, according to the vaccination schedule
Biological: Placebo — Intramuscular dose on Day 42 or on Day -30, according to the vaccination schedule

SUMMARY:
This observer-blind study is designed to evaluate the immune response and safety of pandemic influenza vaccine in the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 61 years or above at the time of the first study visit (Day -30).
* Female subjects of non-childbearing potential.
* Healthy subjects or subjects with well controlled chronic medical condition (at the discretion of the investigator).
* Written informed consent obtained from the subject.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.

Exclusion Criteria:

* Previous administration of the licensed MF59-containing vaccines, e.g. Fluad™ or Addigrip™ or virosome-based influenza vaccines such as Inflexal V™, InfectoVac Flu™ or Invivac™ .
* Previous administration of the 2009 Southern Hemisphere or 2008-2009 Northern Hemisphere influenza vaccine.
* Previous administration of a pandemic influenza vaccine.
* Administration of licensed vaccines within 4 weeks prior to enrolment in this study.
* Planned administration of a vaccine not foreseen by the study protocol up to 30 days after the second vaccination with H5N1 vaccine.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first study vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of chronic alcohol consumption and/or drug abuse.
* History of hypersensitivity to vaccines.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Acute disease and/or fever at the time of enrolment.
* Serious chronic disease including any medically significant chronic pulmonary, cardiovascular, renal, neurological, psychiatric or metabolic disorder, as determined by medical history and physical examination..
* Administration of immunoglobulins and/or any blood products within the three months preceding the first study vaccination or during the study.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days prior to the first vaccination, or planned use during the study period.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Min Age: 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Serum HI antibody titres | Day -30, Day 42

SECONDARY OUTCOMES:
Serum HI antibody titres | Day -30, Day 42, Month 6, Month 12
Serum neutralising antibody titres | Day -30, Day 42, Month 6, Month 12
Occurrence, intensity, and relationship to vaccination of solicited local and general signs and symptoms | Day 0 - Day 6 after each vaccination
Occurrence, intensity and relationship to vaccination of unsolicited adverse events | Day 0 - Day 29 after vaccination, Day 0 - Day 20 after investigational vaccination
Occurrence and relationship to vaccination of serious adverse events | Day 0 - Month 6
Occurrence of adverse events of specific interest | Day 0 - Month 12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Curitiba/Paraná, Paraná, Brazil